CLINICAL TRIAL: NCT05061654
Title: CEFtolozane-Tazobactam for the Empiric Anti-bacterial Treatment of Neutropenic Fever in Hematology Patients; a Single-arm, Single-center, Open-label Clinical Trial (CEF-10 Study)
Brief Title: CEFtolozane-Tazobactam for the Empiric Anti-bacterial Treatment of Neutropenic Fever in Hematology Patients
Acronym: CEF-10
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Administrative constraints
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRC-02-21-015
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2021-09

CONDITIONS: Neutropenia, Febrile; Hematologic Cancer
MeSH Terms: conditions — Febrile Neutropenia; Hematologic Neoplasms | interventions — ceftolozane, tazobactam drug combination

STUDY DESIGN:
Intervention Model Description: The study will be a prospective, non-comparative, single-arm, single center, open-label interventional study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment arm (Experimental): Eligible patients will be started on empiric ceftolozane-tazobactam in addition to standard care.
  Interventions: Drug: Ceftolozane-tazobactam IV

INTERVENTIONS:
Drug: Ceftolozane-tazobactam IV — Empiric Ceftolozane-tazobactam IV 3g over 1 hour every 8 hours. The dose will be reduced to 1.5g 8 hourly in patients with CrCl of 30-50 ml/min, and to 750mg every 8 hours in those with CrCl of 15-29 ml/min. Patients on hemodialysis will receive 2.25g loading dose followed by 450mg every 8 hours.
  Other Names: Zerbaxa

SUMMARY:
Patients with blood cancers and those who received a bone marrow transplant frequently have low circulating white blood cell countS. Fever in patients with low white blood cell count requires early appropriate antibiotic treatment to prevent complications including death. Bacteria have increasingly become more resistant to existing antibiotic options. Ceftolozane-tazobactam is a newer type of antibiotic that has been shown to be safe and effective in infections caused by several types of resistant bacteria that can cause serious infections in individuals with low blood count. This study aims to examine the effectiveness of this antibiotic in these types of patients.

Patients with blood cancer and those who have received a bone transplant will be offered the option to join this study if they develop unexplained fever. If informed consent is granted, they will receive ceftolozane-tazobactam on top of the usual care that such patients receive. The patients will then be followed very closely to check their response to the treatment and if they develop any untoward events. The study will include 164 patients over an estimated 2 year period.

The study is funded by Merck & Co, the company that manufactures the study antibiotic. However, Merck & Co. will not be involved in the actual running of the study, the collection of the study results or their analysis and interpretation. The study protocol has been reviewed and approved by an independent research oversight committee.

DETAILED DESCRIPTION:
The role of early appropriate empiric anti-bacterial therapy in reducing morbidity and mortality in patients with prolonged neutropenia has long being documented. The National Center for Cancer Care and Research (NCCCR) antibiograms for recent years showed increasing rates of ESBL-producing E. coli and K. pneumoniae, as well as reduced susceptibility of P. aeruginosa isolates to piperacillin-tazobactam. Ceftolozane-tazobactam is a newer β-lactam-β-lactamase inhibitor combination with a broad in-vitro spectrum that includes ESBL and AmpC-producing Enterobacterales, as well as multidrug resistant P. aeruginosa. The clinical efficacy and safety of ceftolozane-tazobactam was demonstrated in registrational randomized clinical trials in multiple settings. However, clinical experience with ceftolozane-tazobactam in patients with hematological malignancy or HSCT is very limited. The aim of this study is to explore the potential role of ceftolozane-tazobactam as empiric treatment for hematology patients with neutropenic fever of unknown origin.

The primary objective is to assess the efficacy of ceftolozane-tazobactam as empiric anti-bacterial therapy for neutropenic fever in patients with hematological malignancy or HSCT.

The study will be a prospective, non-comparative, single-arm, single center, open-label interventional study. Patients admitted to NCCCR with a malignant hematological diagnosis and/or HSCT will be screened daily for possible inclusion in the study. Participants will receive empiric therapy with ceftolozane-tazobactam intravenously. All remaining care will be consistent with standard clinical care for patients with neutropenic fever. The Primary endpoint will be treatment success at 72 hours of ceftolozane-tazobactam therapy without modification of anti-bacterial therapy. Treatment success is defined as a composite of defervescence, resolution of any baseline clinical signs of infection, microbiological eradication of any baseline bacterial pathogen, and no modification of anti-bacterial therapy by addition of or switch to an agent with microbiological activity against Enterobacterales or P. aeruginosa (except the addition of sulfamethoxazole-trimethoprim for P. jiroveci prophylaxis).

The study will be conducted in full conformance with principles of the "Declaration of Helsinki", Good Clinical Practice (GCP), and within the laws and regulations of Ministry of Public Health in Qatar. Participation will be subject to written informed consent. The study is sponsored by Hamad Medical Corporation. Funding and medication supply is provided by Merck & Co (MSD) through its Investigator Initiated Studies Program. MSD will not have any role in data collection, data analysis or driving study conclusions.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with an underlying diagnosis of hematological cancer or receipt of hematopoietic stem cell transplantation.
* Age ≥18 years.
* Absolute neutrophil count (ANC) of <0.5x10^9/L or <1.0x10^9/L with a predicted decline to <0.5x10^9/L within the next 2 days.
* Oral temperature of ≥ 38.3 °C once, ≥ 38.0 °C lasting for at least 1 hour, or ≥ 38.0 °C twice within 12 hours.

Exclusion Criteria:

* Allergy to cephalosporins.
* Expected survival of ≤72 hours.
* Expected ANC recovery within ≤72 hours.
* Receipt of any antipseudomonal carbapenem therapy within the preceding 14 days.
* Documented current or past infection or colonization with ceftolozane-tazobactam- resistant Enterobacterales or P. aeruginosa.
* Pregnancy.
* Previous enrollment in CEF-10 Study (subjects previously enrolled in this study cannot be enrolled again during subsequent episodes of neutropenic fever).
* Ongoing therapy or planned continuation of therapy outside the National Center for Cancer Care and Research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Treatment success without modification of anti-bacterial therapy | 72 hours
  Treatment success is defined as a composite of defervescence, resolution of any baseline clinical signs of infection, microbiological eradication of any baseline bacterial pathogen, and no modification of anti-bacterial therapy by addition of or switch to an agent with microbiological activity against Enterobacterales or P. aeruginosa (except the addition of sulfamethoxazole-trimethoprim for P. jiroveci prophylaxis).

SECONDARY OUTCOMES:
Treatment success without modification of anti-bacterial therapy | 7 days
  Treatment success is defined as a composite of defervescence, resolution of any baseline clinical signs of infection, microbiological eradication of any baseline bacterial pathogen, and no modification of anti-bacterial therapy by addition of or switch to an agent with microbiological activity against Enterobacterales or P. aeruginosa (except the addition of sulfamethoxazole-trimethoprim for P. jiroveci prophylaxis)
Days to defervescence | 30 days
  Counted from the first oral temperature of <38oC which is sustained for ≥48 hours
30-day survival | 30 days
  Survival for 30 days from initiation of therapy

OTHER OUTCOMES:
In-vitro susceptibility to ceftolozane-tazobactam of any Enterobacterales or P. aeruginosa isolated from the study subjects | 30 days
  CLSI breakpoints

CONTACTS AND LOCATIONS:
Overall Officials: Ali S. Omrani, FRCP, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, National Center for Cancer Care and Research, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No